CLINICAL TRIAL: NCT07366047
Title: The Safety and Efficacy of Autologous Probiotics in Patients With Defunctioning Ileostomy Following Low Anterior Resection for Rectal Cancer.
Brief Title: Autologous Probiotics in Patients With Defunctioning Ileostomy Following LAR for Rectal Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Lin Wang, surgeon-in-charge, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: A-PILLAR
Record Dates: First submitted 2026-01-18; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-07

CONDITIONS: Rectal Cancer; Gut Microbiomes; Autologous Probiotic Transplantation; Defunctioning Ileostomy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous Probiotics Transplantation (Experimental): Patients with defunctioning ileostomy following low anterior resection for rectal cancer, receive autologous probiotic (lactobacillus and bifidobacterium) after ileostomy closure.
  Interventions: Dietary Supplement: Autologous Probiotics

INTERVENTIONS:
Dietary Supplement: Autologous Probiotics — Patients with defunctioning ileostomy following low anterior resection for rectal cancer, receive autologous probiotics (lactobacillus and bifidobacterium) after ileostomy closure.
  All patients will take a 100-day supply of high-activity autologous probiotic enteric-coated capsules (100 lactobacillus and 100 bifidobacterium enteric-coated capsules, 1 capsule per day, with each capsule containing a CFU activity of no less than 100 billion)

SUMMARY:
Rectal cancer patients who received low anterior resection combined with ileostomy may effectively reduce the probability of anastomotic leakage after surgery. However, due to the long-term semi-abandoned state of the distal colon, the probability of bowel dysfunction after ileostomy closure is very high. The incidence of low anterior resection syndrome (LARS) exceeds 70%, which is twice that of those who did not receive a preventive stoma. The main reasons include postoperative anatomical structure alteration, nerve damage, pathological changes of the colorectal mucosa, and gut microbiota variation, etc. The application of probiotics can significantly improve the bowel function of these patients. In this study, in order to enhance the colonization effect of probiotics, autologous probiotics will be applied to treat patients with defunctioning ileostomy. The primary outcome is the occurrence of major LARS after 6 months of the treatment.

DETAILED DESCRIPTION:
The number of new cases and deaths of colorectal cancer in China is increasing year by year, seriously threatening the lives and health of the Chinese people. The incidence of rectal cancer accounts for 70% of colorectal cancer. Among them, patients with low rectal cancer involve the issue of preserving the anal sphincter. In recent years, with the improvement of chemoradiotherapy, the organ preservation rate has gradually increased. However, patients with advanced rectal cancer who receive neoadjuvant chemoradiotherapy usually need to undergo an ileostomy to decrease the rate of leakage. After ileostomy closure, patients may experience various adverse reactions such as intestinal obstruction, diarrhea, and constipation. The incidence of low anterior resection syndrome (LARS) exceeds 70%. Normally, the distal colon of patients with an ileostomy is in a semi-abandoned state for a long time. The composition of gut microbiota is significantly different, which is an important factor in leading to LARS. Therefore, the regulation of gut microbiota plays an important role in the recovery of bowel function in these patients.

The human body is a complex symbiotic life form composed of its own cells and a large number of symbiotic microbial cells. The number of microorganisms in the human gastrointestinal tract is ten times the number of human cells; the number of genes contained in microorganisms exceeds 10 million, which is 150 times the number of human genes. Gut bacteria have multiple functions, such as food fermentation, protecting the human body from pathogens, stimulating immune responses, and producing vitamins. At the same time, gut microbiota is involved in many kinds of bowel disease. The regulation of gut microbiota composition in the gut is a useful therapeutic strategy for bowel disease. Fecal microbiota transplantation (FMT) is defined as transplanting the functional microbiota from the feces of a healthy person into the gastrointestinal tract of a patient to restore the patient's normal intestinal microbiota and thereby improve intestinal function and overall health. It is divided into autologous fecal microbiota transplantation (aFMT) and heterologous fecal microbiota transplantation (hFMT). Normally, aFMT can improve the restoration of gut microbiota compared with the method of hFMT. Some kinds of disease should be treated by restoring the gut microbiota environment with autologous probiotics to enhance immunity and prevent the possibility of disease occurrence.

This study is a single-arm, single-center clinical trial, and it plans to include 40 rectal cancer patients with ileostomy. Patients with an ileostomy received autologous probiotics (lactobacillus and bifidobacterium) after the ileostomy closure. All patients will take a 100-day supply of high-activity autologous probiotic enteric-coated capsules (100 lactobacillus and 100 bifidobacterium enteric-coated capsules, 1 capsule per day, with each capsule containing a Colony-Forming Units (CFU) activity of no less than 100 billion). The primary outcome is the occurrence of major LARS after 6 months of the treatment. The secondary outcome measures, including quality of life impairment, LARS score, bowel function impairment, fecal continence impairment, were detected after ileostomy closure (1, 3, 6, 12 months). in order to provide new ideas for the treatment of LARS, the aim of this study is to observe the safety and efficacy of autologous probiotics in patients with ileostomy closure and to investigate improvement on LARS in these patients.

ELIGIBILITY:
Inclusion Criteria:

Age: 18-80years old; Curative low anterior resection for rectal cancer with defunctioning ileostomy; ileostomy closure within 3-6 month; Preoperative chemoradiotherapy ; No evidence of anastomotic leakage or severe stenosis

Exclusion Criteria:

Tumor recurrence or distant metastasis; Secondary operation with stoma; Prior disease impairing bowel function except for rectal cancer; Any contraindication for transanal irrigation; Pregnant or nursing; Serious cardiovascular disease, uncontrolled infections, or other serious uncontrolled concomitant disease; Cognitive or psychological disorder;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with major low anterior resection syndrome score (LARS score) | at the time of 6 months since the start of treatment

SECONDARY OUTCOMES:
Quality of life impairment assessed by Short Form 36 (SF-36) | at the time of 1, 3, 6, 12 months since the start of treatment
  Quality of life will be assessed by Short Form 36 (SF-36) health questionnaire.
Number of participants with major low anterior resection syndrome score (LARS score) | at the time of1, 3, 6, 12months since the start of treatment
Bowel function impairment | at the time of 1, 3, 6, 12 months since the start of treatment
  Bowel function will be assessed by Memorial Sloan Kettering Cancer Centre Bowel Function Instrument (MSKCC BFI). Stool frequency will be recorded in the day and night.
Fecal continence impairment | at the time of 6, 12 months since the start of treatment
  Fecal incontinence will be assessed by Wexner incontinence scale (WIS).

IPD SHARING:
Plan to Share IPD: Undecided